CLINICAL TRIAL: NCT00800800
Title: Effect of Cholesterol Lowering on the Progression of Aortic Stenosis in Patients With Mild to Moderate Aortic Stenosis (ASTRONOMER)Aortic Stenosis Progression Observation Measuring Effects of Rosuvastatin and The Sub-Study Protocol.
Brief Title: Effects of Rosuvastatin on Aortic Stenosis Progression
Acronym: ASTRONOMER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Andrew Vieira, AstraZeneca Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DC-452-0003
Record Dates: First submitted 2008-11-25; First posted 2008-12-02 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Aortic Stenosis
Keywords: progression of aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rosuvastatin 40 mg
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg, oral, single dose
  Arms: 1
Drug: Placebo — oral, single dose
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effects of rosuvastatin compared to usual care in patients diagnosed with aortic valvular stenosis. Patients must have a diagnosis of mild to moderate aortic stenosis (AS) and no clinical indication for the use of cholesterol lowering agents. A multi-centre, randomized, double-blind, placebo-controlled study, with a two year recruitment period, and a treatment duration of a minimum of 3 years from the time of the last patient randomized to a maximum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate AS defined by peak Doppler aortic valve velocity 2.5 to 4 m/sec
* Baseline LDL-C value must be within targeted level for all risk categories according to the Canadian Guidelines
* Baseline triglyceride levels must be within target level for the risk categories

Exclusion Criteria:

* Very mild AS defined by peak Doppler AS velocity <2.5m/sec, because the rate of progression is not well defined; Females of child bearing potential who do not practice adequate contraception.
* Severe AS defined by peak Doppler AS velocity > 4m/sec. These patients are excluded because they will have a high probability of aortic valve replacement even without further AS progression.
* Greater than moderate aortic regurgitation, defined as aortic jet width to aortic outflow tract ratio >0.45; Patients with diabetes or with a fasting blood sugar level > 7.0 mmol/L (must be confirmed with one repeat assay within 14 days).
* Significant concomitant mitral valve disease, defined by > moderate mitral regurgitation (MR) or mitral valve area (MVA)< 1.5 cm2; A very high risk of CAD (10 year risk > 30%), according to the Canadian Guidelines.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2002-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The changes in transvalvular aortic velocities and the changes in aortic valve area. | Between baseline and close-out measurments.

SECONDARY OUTCOMES:
The incidence and severity of adverse events, the clinically relevant changes in echocardiograms, and laboratory analysis will be compared between the two treatment groups. | Baseline and minimum of 3 year follow-up.
The incidence and severity of adverse events, the clinically relevant changes in echocardiograms, and laboratory analysis will be compared between the two treatment groups. | Between baseline and close-out measurments.

CONTACTS AND LOCATIONS:
Locations (15):
- Canada (15):
  - Research site, Calgary, Alberta
  - Research site, Edmonton, Alberta
  - Research site, Surrey, British Columbia
  - Research site, Vancouver, British Columbia
  - Research site, Victoria, British Columbia
  - Research site, Edmonton, Manitoba
  - Research site, Brampton, Ontario
  - Research site, Cambridge, Ontario
  - Research site, Kitchener, Ontario
  - Research site, Montreal, Ontario
  - Research site, Ottawa, Ontario
  - Research site, Toronto, Ontario
  - Research site, Montreal, Quebec
  - Research site, Halifax
  - Research site, St. John's

REFERENCES:
- [Derived] Capoulade R, Torzewski M, Mayr M, Chan KL, Mathieu P, Bosse Y, Dumesnil JG, Tam J, Teo KK, Burnap SA, Schmid J, Gobel N, Franke UFW, Sanchez A, Witztum JL, Yang X, Yeang C, Arsenault B, Despres JP, Pibarot P, Tsimikas S. ApoCIII-Lp(a) complexes in conjunction with Lp(a)-OxPL predict rapid progression of aortic stenosis. Heart. 2020 May;106(10):738-745. doi: 10.1136/heartjnl-2019-315840. Epub 2020 Feb 13. PMID 32054669
- [Derived] Capoulade R, Yeang C, Chan KL, Pibarot P, Tsimikas S. Association of Mild to Moderate Aortic Valve Stenosis Progression With Higher Lipoprotein(a) and Oxidized Phospholipid Levels: Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2018 Dec 1;3(12):1212-1217. doi: 10.1001/jamacardio.2018.3798. PMID 30476957
- [Derived] Capoulade R, Chan KL, Mathieu P, Bosse Y, Dumesnil JG, Tam JW, Teo KK, Yang X, Witztum JL, Arsenault BJ, Despres JP, Pibarot P, Tsimikas S. Autoantibodies and immune complexes to oxidation-specific epitopes and progression of aortic stenosis: Results from the ASTRONOMER trial. Atherosclerosis. 2017 May;260:1-7. doi: 10.1016/j.atherosclerosis.2017.03.013. Epub 2017 Mar 9. PMID 28319871
- [Derived] Capoulade R, Chan KL, Yeang C, Mathieu P, Bosse Y, Dumesnil JG, Tam JW, Teo KK, Mahmut A, Yang X, Witztum JL, Arsenault BJ, Despres JP, Pibarot P, Tsimikas S. Oxidized Phospholipids, Lipoprotein(a), and Progression of Calcific Aortic Valve Stenosis. J Am Coll Cardiol. 2015 Sep 15;66(11):1236-1246. doi: 10.1016/j.jacc.2015.07.020. PMID 26361154
- [Derived] Page A, Dumesnil JG, Clavel MA, Chan KL, Teo KK, Tam JW, Mathieu P, Despres JP, Pibarot P; ASTRONOMER Investigators. Metabolic syndrome is associated with more pronounced impairment of left ventricle geometry and function in patients with calcific aortic stenosis: a substudy of the ASTRONOMER (Aortic Stenosis Progression Observation Measuring Effects of Rosuvastatin). J Am Coll Cardiol. 2010 Apr 27;55(17):1867-74. doi: 10.1016/j.jacc.2009.11.083. PMID 20413039